CLINICAL TRIAL: NCT02930486
Title: Ziptight or Tricortical Screw Fixation of Acute Tibiofibular Syndesmotic Injury
Acronym: S16
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other); Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Syndesmose2016
Record Dates: First submitted 2016-04-18; First posted 2016-10-12 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Ankle Fractures
Keywords: Syndesmosis; Injury; Ankle; Fracture; Weber C
MeSH Terms: conditions — Ankle Fractures; Wounds and Injuries; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZipTight (Active Comparator): ZipTight suture endobutton
  Interventions: Device: ZipTight suture endobutton
- Syndesmotic screw (Active Comparator): Tricortical 3.5 mm syndesmotic screw
  Interventions: Device: Tricortical 3.5 mm syndesmotic screw

INTERVENTIONS:
Device: ZipTight suture endobutton — Zimmer Biomet ZipTight suture endobutton
  Arms: ZipTight
Device: Tricortical 3.5 mm syndesmotic screw — Depuy Synthes 3.5 mm screw
  Arms: Syndesmotic screw

SUMMARY:
Treatment of syndesmotic injury with Weber C fracture. A randomized study comparing ZipTight suture endobutton and one tricortical 3,5 mm syndesmotic screw.

DETAILED DESCRIPTION:
Syndesmotic injuries are common and often associated with unstable ankle fractures. The most common treatment is with a syndesmotic screw through the fibula and tibia which is later removed, usually after 10-12 weeks. The ZipTight suture endobutton (Biomet) is used for the same indication. It does not need removal and thus avoids subsequent surgery. This trial will compare these two methods and see if they are equal.

patients 18-70 years presenting to one of the three hospitals with and acute syndesmotic injury are eligible for inclusion. 120 patients are randomized to two treatment groups. One group will be treated with a ZipTight suture endobutton fixation and the other receives a tricortical screw fixation. Neither suture endobutton or screw is routinely removed. Follow up intervals are at 6 weeks, 6, 12 and 24 months with clinical and-points. Standardized CT scans are taken postoperatively and at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years
* Acute syndesmotic injury with Weber type C fracture

Exclusion Criteria:

* Prior injury og the same ankle
* Severe injury of the same leg affecting rehabilitation
* Symptomatic osteoarthritis of same ankle
* open injury
* Decubital injury affecting surgical site
* Dementia or unable to sign informed consent
* neuropatic conditions affecting same leg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01; Primary Completion 2017-09-30 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
OTA Score (Modified American Orthopaedic Foot and Ankle Society ankle hind foot score) | 24 months
  Modified American Orthopaedic Foot and Ankle Society ankle hind foot score (0-100)

SECONDARY OUTCOMES:
Manchester-Oxford Foot questionnaire (MOxFQ) | 24 months
Dorsiflexion angle | 24 months
  according to Lindsjø
Health-related quality of life (EQ-5D) | 24 months
CT measurements of syndesmotic distance | 24 months
VAS | 24 months
  visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Baerum Hospital, Vestre Viken, Sandvika, Gjettum, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raeder BW, Stake IK, Madsen JE, Frihagen F, Jacobsen SB, Andersen MR, Figved W. Randomized trial comparing suture button with single 3.5 mm syndesmotic screw for ankle syndesmosis injury: similar results at 2 years. Acta Orthop. 2020 Dec;91(6):770-775. doi: 10.1080/17453674.2020.1818175. Epub 2020 Sep 10. PMID 32907456